CLINICAL TRIAL: NCT01887743
Title: The Effect of Obesity on the Pharmacokinetics of Pantoprazole and CYP2C19 Activity in Children and Adolescents With GERD
Brief Title: Pharmacokinetics of Pantoprazole and CYP2C19 Activity in Children and Adolescents With GERD: A Pilot Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: G130069PTZ-BT
Record Dates: First submitted 2013-06-19; First posted 2013-06-27 (Estimated); Results first posted 2021-12-03 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-10

CONDITIONS: Obesity; GERD
Keywords: GERD; Obesity; Pediatric; Pantoprazole; CYP2C19; Pharmacokinetic
MeSH Terms: conditions — Obesity; Gastroesophageal Reflux | interventions — Pantoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pantoprazole (Experimental): This will be a single dose study where participants will receive 1.2mg/kg or no more than 100mg total one time dose as a liquid containing Carbon 13 labeled Pantoprazole with a final concentration of 4.0mg/mL.
  Interventions: Drug: Pantoprazole

INTERVENTIONS:
Drug: Pantoprazole — This will be a single dose study where participants will receive 1.2mg/kg or no more than 100mg total one time dose as a liquid containing Carbon 13 labeled Pantoprazole with a final concentration of 4.0mg/mL.
  Other Names: Protonix

SUMMARY:
The World Health Organization has declared childhood obesity to be "one of the most serious public health challenges of the 21st century," (http://www.who.int/dietphysicalactivity/childhood). Given that obese children are generally excluded from clinical trials, little to no information exists regarding the impact of obesity on drug disposition and drug action, creating a gap in physicians' knowledge on how to appropriately select the dose of many critical medications (e.g., anticancer agents), so as to prevent toxicity associated with overdosing, while avoiding the harms of under-treatment. The proposed study will examine the effect of obesity on the metabolism of a commonly used medication, the proton pump inhibitor pantoprazole, by exploring the relationships between age, obesity, basal metabolic rate and genetic control of the enzyme primarily responsible for pantoprazole metabolism. We will also validate a simple breath test that can be used to predict pantoprazole dose requirement for obese children.

The study is designed to test the following experimental hypotheses:[13C]-pantoprazole pharmacokinetic parameters are not different between non-obese and obese children and adolescents, collectively (both age groups combined) or stratified by age group (SA 1) [13C]-pantoprazole pharmacokinetic parameters or DOB values (and thus, CYP2C19 activity) are not different between males and females (SA 1 & 2) [13C]-pantoprazole pharmacokinetic parameters and DOB (Delta over baseline) values (and thus, CYP2C19 activity) are independent of age over the age range of 6 to 17 years (SA 1 & 2) Obesity does not alter the relative contributions of CYP2C19-dependent and non-CYP2C19-dependent (i.e., CYP3A4) metabolism of pantoprazole, as measured by the urinary ratio of 4-hydroxy-pantoprazole to pantoprazole sulfone (SA 1 & 2) The [13C]-pantoprazole breath test, by determining DOB at discrete time point(s), is a non-invasive measure of CYP2C19 phenotype (SA 2) Clearance of pantoprazole (surrogate for CYP2C19 activity) is a function of REE in obese and non-obese children and adolescents (SA 3) Pantoprazole clearance (surrogate for CYP2C19 activity) is associated with fat distribution, as determined by waist-to-hip ratios (SA 3)

DETAILED DESCRIPTION:
As the pediatric obesity epidemic continues to rise, obesity-associated pathologic conditions, such as type II diabetes, hypertension and gastroesophageal reflux disease (GERD), become more prevalent, which, in turn, creates a need for a better understanding of the impact of obesity on drug disposition and response in pediatric patients with obesity. The following proposal is designed to address the hypothesis that obesity per se has significant effects on the pharmacokinetics of CYP2C19 substrates in children and adolescents. Pantoprazole, a proton pump inhibitor (PPI) frequently used in the treatment of GERD and related conditions, is ideally suited for such a study, given the predominant role of CYP2C19(Cytochrome P450 subtype 2C19) in its metabolism and its favorable safety and efficacy profile in pediatric medicine. The study of obesity on the activity of CYP2C19 is relevant, as it has not been previously studied in pediatrics and the enzyme catalyzes the biotransformation of over 20 drugs frequently used in pediatrics (eg., PPIs, selective serotonin re-uptake inhibitors). Moreover, knowledge of the CYP2C19 genotype and phenotype can be used to individualize drug treatment, making treatment safer and more effective for children. The primary objective of the proposed investigation is to evaluate the effect of obesity on the pharmacokinetics of pantoprazole in children and adolescents. The secondary objective is to assess the utility of the [13C]-pantoprazole breath test, a novel, non-invasive, in-vivo technique, as a surrogate biomarker of CYP2C19 activity in pediatric patients. In addition, the impact of non-genetic variables, such as resting energy expenditure (REE), on CYP2C19 activity will be investigated. The proposed research objectives will be achieved by administration of a single dose of oral [13C]-pantoprazole, a safe and stable non-radioactive isotope, to 100 patients (both male and female), including 50 obese (as defined by BMI >95th percentile) and 50 non-obese patients, between the ages of 6-17 years. Breath samples will be collected before, and for 8 hours after, [13C]-pantoprazole administration to quantify 13CO2(Carbon 13 dioxide)/12CO2(Carbon 12 dioxide) by infrared spectrometry. Simultaneously, repeated blood sampling will be used to measure pantoprazole, and its primary CYP2C19 catalyzed metabolite. Pantoprazole disposition will then be characterized from both breath sample and plasma level data and examined in association with important covariates (e.g., age, hip:waist ratio, BMI, REE, parent drug:metabolite ratio and CYP2C19 genotype) to test the experimental hypothesis. Data will be collected and analyzed by a team of highly experienced investigators representing the fields of gastroenterology, pediatric clinical pharmacology and the evolving field of obesity medicine.

ELIGIBILITY:
Inclusion Criteria

* Males and females between 6 and 17 years of age.
* Pediatric patients who have a primary diagnosis of GERD or related symptoms, defined as one or more of the following: clinical symptoms consistent with GERD, a diagnosis of erosive esophagitis by endoscopy, esophageal biopsy with histopathology consistent with reflux esophagitis, abnormal pH probe study consistent with reflux esophagitis, or other test result consistent with GERD.
* Non-obese: 10th - 84th percentile for BMI (50 subjects)
* Overweight: greater than 85th percentile for BMI (50 subjects)
* Provide written assent with parental permission

Exclusion Criteria

* Inability to have blood drawn for the screening lab tests
* Current therapy with medications known to clinically significantly inhibit or to induce CYP2C19, such as phenytoin, oxcarbazepine, carbamazepine, and rifampicin
* Inability or unwillingness to fast overnight prior to the study session
* Established diagnosis of asthma with evidence of an exacerbation < 5 days before administration of the study article. Children with asthma that is well controlled on maintenance treatment will be eligible for enrollment to the study
* Existence of metabolic disease
* A demonstrated adverse reaction to previous pantoprazole or PPI exposure
* Impaired hepatic activity as determined by routine liver function testing and defined as values greater than or equal to 3 times the age-specific upper limit of normal (ULN) for AST(aspartate amino transferase), ALT (alanine amino transferase), total bilirubin >2.0 mg/dl, alkaline phosphatase greater than or equal to 5 times the age-specific ULN
* Impaired renal function defined as greater than or equal to 3 times the age-specific ULN
* For females, a positive urine beta-human chorionic gonadotropin pregnancy test result
* Any known infection with hepatitis B, C, or human immunodeficiency virus (HIV)

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 71 (Actual)
Dates: Start 2013-06; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Friesen, MD, Principal Investigator — Children's Mercy Hospital and Clinics
Locations (1):
- Children's Mercy Hospital and Clinics, Kansas City, Missouri, United States

REFERENCES:
- [Derived] Shakhnovich V, Abdel-Rahman S, Friesen CA, Weigel J, Pearce RE, Gaedigk A, Leeder JS, Kearns GL. Lean body weight dosing avoids excessive systemic exposure to proton pump inhibitors for children with obesity. Pediatr Obes. 2019 Jan;14(1):10.1111/ijpo.12459. doi: 10.1111/ijpo.12459. Epub 2018 Sep 26. PMID 30257076

RESULTS

PARTICIPANT FLOW:
Groups:
- Obese: BMI for age at or above the 95th percentile
- Overweight: BMI for age 85-94th percentile
- Normal Weight: BMI for age <85th percentile
Period: Overall Study
Arm/Group | Obese | Overweight | Normal Weight
Started | 20 | 19 | 32
Completed | 19 | 17 | 29
Not Completed | 1 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Normal Weight: BMI10-84th percentile for age
- Overweight: BMI 85-94th percentile for age
- Obese: BMI at or above 95th percentile for age
- Total: Total of all reporting groups
Arm/Group | Normal Weight | Overweight | Obese | Total
Number analyzed (Participants) | 29 | 17 | 19 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.7 (3.8) | 14.9 (2.6) | 12.7 (3.0) | 13.7 (3.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 13 | 40
  Male | 15 | 4 | 6 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 4 | 6
  Not Hispanic or Latino | 27 | 17 | 15 | 59
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 29 | 17 | 17 | 63
BMI percentile for age [Mean (Standard Deviation); unit: percentile for age] | 62.0 (18.2) | 89.3 (2.5) | 97.7 (1.8) | 79.0 (19.9)

OUTCOME MEASURES:

1. Primary Outcome: Pantoprazole Apparent Oral Clearance
Description: Pantoprazole apparent oral drug clearance (CL/F) adjusted for weight for children with the most common CYP2C19 genotypes (i.e., *1/1, *1/17, *1/2, *2/17). Only children with evaluable plasma samples (i.e., at least 85% of planned plasma samples collected) were included in this analysis (n=57).
Time Frame: 8 hours
Population: Only children with evaluable plasma samples (i.e., at least 85% of planned plasma samples collected) were included in this analysis (n=57).
Measure: Mean (Standard Deviation); unit: L/hr/kg
Arm/Group | Normal Weight | Overweight | Obese
Number analyzed (Participants) | 28 | 16 | 13
L/hr/kg | 0.42 (0.27) | 0.29 (0.12) | 0.23 (0.13)

2. Primary Outcome: Unadjusted Pantoprazole Apparent Oral Clearance
Description: Pantoprazole apparent oral drug clearance (CL/F), not adjusted for weight, for children with the most common CYP2C19 genotypes (i.e., *1/1, *1/17, *1/2, *2/17). Only children with evaluable plasma samples (i.e., at least 85% of planned plasma samples collected) were included in this analysis (n=57).
Time Frame: 8 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Normal Weight | Overweight | Obese
Number analyzed (Participants) | 28 | 16 | 13
L/hr | 20.4 (14.2) | 18.7 (7.43) | 16.8 (8.55)

3. Secondary Outcome: Precision of Breath Test to Discriminate the CYP2C19 Extensive Metabolizer (EM) From Intermediate Metabolizer (IM) Phenotype
Description: Children with common CYP2C19 genotypes (*1/*1, *1*17, *1/*2, *2/*17) who had evaluable breath test data (n=59) were included to evaluate the breath test's precision in discriminating the CYP2C19 Extensive Metabolizer (EM; *1/*1, *1*17) from the Intermediate Metabolizer (IM; *1/*2, *2/*17) phenotype in the first 3 hrs after study drug administration. A 3-hour window was chosen for convenience. A predictive model using breath test features (change in ratio of C12-to-C13 in exhaled CO2) was build and validated to predictphenotype for each child. We drew bootstrap samples, each stratified to preserve the observed prevalence of EM/IMs in the original cohort (n=59). Sampling with replacement left out 38% of the original sample to use as a test dataset to validate model performance. For each bootstrap sample, a 500-tree Extremely randomized Extra-Tree Forest was constructed after seeding. Using phenotypes predicted by the forest, predictive accuracy was assessed by computing precision.
Time Frame: 3 hours
Population: The mean precision was calculated at 5 timepoints during the first 3 hours post-drug administration to test the breath test's ability to discriminate CYP2C19 EM from IM. All EM/IM children with evaluable breath test data were included as a single study group in this analysis.
Measure: Mean (Standard Deviation); unit: percent true EM in total EM predicted
Groups:
- Breath Test: Children with evaluable breath data and the following CYP2C19 genotypes *1/*1, *1/17 (i.e., extensive metabolizer) and *1/*2 ,*2/*17 (i.e., intermediate metabolizer) were included in the breath test analyses (n=59) to assess how well the test could discriminate CYP2C19 extensive metablizers (EM) from intermediate metabolizers (IM).
Arm/Group | Breath Test
Number analyzed (Participants) | 59
percent true EM in total EM predicted
  30 minutes | 77.3 (5.5)
  60 minutes | 77.7 (5.0)
  90 minutes | 77.3 (5.0)
  120 minutes | 77.8 (5.1)
  180 minutes | 76.9 (5.0)

4. Secondary Outcome: Recall of Breath Test to Discriminate the CYP2C19 Extensive Metabolizer (EM) From Intermediate Metabolizer (IM) Phenotype
Description: Children with common CYP2C19 genotypes (*1/*1, *1*17, *1/*2, *2/*17) who had evaluable breath test data (n=59) were included to evaluate the breath test's precision in discriminating the CYP2C19 Extensive Metabolizer (EM; *1/*1, *1*17) from the Intermediate Metabolizer (IM; *1/*2, *2/*17) phenotype in the first 3 hrs after study drug administration. A 3-hour window was chosen for convenience. A predictive model using breath test features (change in ratio of C12-to-C13 in exhaled CO2) was build and validated to predictphenotype for each child. We drew bootstrap samples, each stratified to preserve the observed prevalence of EM/IMs in the original cohort (n=59). Sampling with replacement left out 38% of the original sample to use as a test dataset to validate model performance. For each bootstrap sample, a 500-tree Extremely randomized Extra-Tree Forest was constructed after seeding. Using phenotypes predicted by the forest, predictive accuracy was assessed by computing recall.
Time Frame: 3 hours
Population: The mean recall was calculated at 5 timepoints during the first 3 hours post-drug administration to test the breath test's ability to discriminate CYP2C19 EM from IM. All EM/IM children with evaluable breath test data were included as a single study group in this analysis.
Measure: Mean (Standard Deviation); unit: percent identified EM out of total EM
Arm/Group | Breath Test
Number analyzed (Participants) | 59
percent identified EM out of total EM
  30 minutes | 87.8 (9.5)
  60 minutes | 93.6 (7.9)
  90 minutes | 92.3 (7.9)
  120 minutes | 92.4 (7.5)
  180 minutes | 90.2 (8.1)

5. Secondary Outcome: Harmonic Mean of Precision and Recall (F1) of the Breath Test to Discriminate the CYP2C19 Extensive Metabolizer (EM) From Intermediate Metabolizer (IM) Phenotype
Description: Children with common CYP2C19 genotypes (*1/*1, *1*17, *1/*2, *2/*17) who had evaluable breath test data (n=59) were included to evaluate the breath test's precision in discriminating the CYP2C19 Extensive Metabolizer (EM; *1/*1, *1*17) from the Intermediate Metabolizer (IM; *1/*2, *2/*17) phenotype in the first 3 hrs after study drug administration. A 3-hour window was chosen for convenience. A predictive model using breath test features (change in ratio of C12-to-C13 in exhaled CO2) was build and validated to predictphenotype for each child. We drew bootstrap samples, each stratified to preserve the observed prevalence of EM/IMs in the original cohort (n=59). Sampling with replacement left out 38% of the original sample to use as a test dataset to validate model performance. For each bootstrap sample, a 500-tree Extremely randomized Extra-Tree Forest was constructed after seeding. Using phenotypes predicted by the forest, predictive accuracy was assessed by computing the F1.
Time Frame: 3 hours
Population: The mean F1 was calculated at 5 timepoints during the first 3 hours post-drug administration to test the breath test's ability to discriminate CYP2C19 EM from IM. All EM/IM children with evaluable breath test data were included as a single study group in this analysis.
Measure: Mean (Standard Deviation); unit: percent mean predictive performance
Arm/Group | Breath Test
Number analyzed (Participants) | 59
percent mean predictive performance
  30 minutes | 81.9 (5.5)
  60 minutes | 84.7 (4.7)
  90 minutes | 83.8 (4.6)
  120 minutes | 84.3 (4.5)
  180 minutes | 82.8 (4.7)

ADVERSE EVENTS:
Time Frame: 8 hours during the PK study
Arm/Group | Normal Weight | Overweight | Obese
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/19 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 0/32 | 0/19 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes